CLINICAL TRIAL: NCT00651989
Title: Agreement in Foveal Thickness Measurements Between Spectralis® and Stratus® Optical Coherence Tomography
Brief Title: Agreement Between Spectral Domain and Time Domain Optical Coherence Tomography (OCT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Paolo Carpineto M.D., Dept. of Medicine and Aging Sciences, University "G. d'Annunzio" Chieti-Pescara
Other Study IDs: Ud'A-Ophtha-001
Record Dates: First submitted 2008-03-28; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-03

CONDITIONS: Normal Foveal Thickness
Keywords: optical coherence tomography; spectral domain; time domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: healthy individuals
  Interventions: Other: optical coherence tomography foveal thickness measurement

INTERVENTIONS:
Other: optical coherence tomography foveal thickness measurement — In the same session in one randomly selected eye of each subject three consecutive measurements of foveal thickness were performed using both time-domain OCT and spectral-domain OCT.
  Other Names: healthy subjects

SUMMARY:
Optical coherence tomography (OCT) is a well-established and safe technique that offers the possibility of visualizing retinal structure and measuring retinal thickness. Time-domain (TD)OCT is considered the "gold standard" technique for retinal thickness measurements. Spectral-domain (SD) OCT has to face the gold standard technique prior to obtain scientific and clinical consensus.

In our study in healthy subjects foveal thickness will be measured with both TD and SD OCT , and the data will be compared to evidence any difference between the two retinal measurements techniques.

DETAILED DESCRIPTION:
The study will be performed at the Ophthalmology Clinic of the University of Chieti-Pescara, Italy. Forty healthy individuals will be enrolled in this study. In the same session in one randomly selected eye of each subject three consecutive measurements of foveal thickness will be performed using both TD OCT and FD OCT. All measurements will be obtained by the same experienced examinator.

Time domain optical coherence tomography images will be obtained from each eye after pupil dilation using the Stratus OCT system (version 4.1. Carl Zeiss Meditec, Dublin, CA).

Spectral domain optical coherence tomography images will be obtained using the HRA-OCT Spectralis unit (Heidelberg Engineering GmbH, Heidelberg, Germany).

All data will be analyzed with the statistical package MedCalc® version 8.1 for Windows (MedCalc®, Mariakerke, Belgium).

The D'Agostino-Pearson test that computes a single P-value for the combination of the coefficients of Skewness and Kurtosis will be used to study the sample distribution.

T-test will be used to compare means between Stratus and Spectralis measurements and orizontal and vertical measurements.

To assess agreement between Spectralis and Stratus OCT foveal measurements the Bland and Altman plots of the agreement in foveal thickness will be used. For both orizontal and vertical foveal measurements the ratio (Spectralis/stratus OCT foveal thickness) will be plotted against the average of the two measurements.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* any systemic or eye disease
* previous ocular surgery or laser treatment
* any systemic or ocular therapy

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: volounteer students and employers from the Clinic staff
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
foveal thickness | at subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Carpineto, M.D., Principal Investigator — Dept. of Medicine and Aging Sciences, Univ. "G. d'Annunzio" Chieti-Pescara
Locations (1):
- Ophthalmology Clinic, Univ. "G. d'Annunzio" Chieti-Pescara, Chieti, Italy

REFERENCES:
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172